CLINICAL TRIAL: NCT06024746
Title: Combined Efficacy and Safety of an Early, Intensive, Management Strategy with Finerenone and SGLT2 Inhibitor in Patients Hospitalized with Heart Failure (CONFIRMATION-HF)
Brief Title: A Study to Determine the Efficacy and Safety of Finerenone and SGLT2i in Combination in Hospitalized Patients with Heart Failure (CONFIRMATION-HF)
Acronym: CONFIRMATION
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Colorado Prevention Center (Other)
Collaborators: Saint Luke's Mid America Heart Institute (Unknown); Bayer Healthcare Pharmaceuticals, Inc./Bayer Schering Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202303CPC
Record Dates: First submitted 2023-08-22; First posted 2023-09-06 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Heart Failure
Keywords: Heart Failure; Hospitalized
MeSH Terms: conditions — Heart Failure | interventions — finerenone; empagliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Finerenone plus empagliflozin (Experimental)
  Interventions: Drug: Finerenone; Drug: Empagliflozin
- Usual care (No Intervention): Usual care management

INTERVENTIONS:
Drug: Finerenone — Oral finerenone.
  Arms: Finerenone plus empagliflozin
Drug: Empagliflozin — Oral empagliflozin.
  Arms: Finerenone plus empagliflozin

SUMMARY:
Combination therapy of finerenone plus empagliflozin will be compared to usual care to determine the efficacy and safety of treatment in patients hospitalized with heart failure.

DETAILED DESCRIPTION:
This is an international, randomized, controlled, open-label, trial of an early, intensive management strategy using the combination of finerenone plus sodium-glucose co-transporter 2 inhibitor (SGLT2i) compared with usual care in patients hospitalized with heart failure (HF).

ELIGIBILITY:
Inclusion Criteria:

* Provide electronic or written informed consent, either personally or through a legally authorized representative, as permitted by local regulations
* Age ≥18 years or legal age of majority if >18 years in the participant's country of residence
* Current hospitalization or recently discharged with the primary diagnosis of heart failure
* Heart failure signs and symptoms at the time of hospital admission
* Elevated N-terminal pro B-type natriuretic peptide (NTproBNP) ≥500 pg/mL or B-type natriuretic peptide (BNP) ≥125 pg/mL according to the local lab for patients in sinus rhythm; or elevated NTproBNP ≥1500 pg/mL or BNP ≥375 pg/mL for patients with atrial fibrillation (AF), measured during the current hospitalization or in the 72 hours prior to hospital admission
* Fulfillment of protocol defined stabilization criteria (if randomized during hospitalization)
* Treatment during the index hospitalization with at least 1 intravenous dose of a loop diuretic (e.g., furosemide, torsemide, bumetanide).
* Negative pregnancy test and agreement to use adequate contraception during trial (female participants only)

Exclusion Criteria:

* Diagnosis of type 1 diabetes or prior history of diabetic ketoacidosis
* Documented prior history of severe hyperkalemia in the setting of MRA use
* Treatment with non-steroidal mineralocorticoid receptor antagonist (MRA) or SGLT2i
* Estimated glomerular filtration rate (eGFR) <30 mL/min/1.73m² and/or potassium >5.0 mmol/L
* Acute myocardial infarction, coronary revascularization, valve replacement/repair, or implantation of a cardiac resynchronization therapy device within 30 days
* Prior or planned heart transplant
* Hemodynamically significant uncorrected primary cardiac valvular disease as primary cause of heart failure
* Cardiomyopathy due to acute inflammatory heart disease, infiltrative diseases, accumulation diseases, muscular dystrophies, cardiomyopathy with reversible causes, known hypertrophic obstructive cardiomyopathy, complex congenital heart disease, or pericardial constriction
* Probable alternative cause of participant's heart failure symptoms
* Concomitant systemic therapy with potent cytochrome P450 isoenzyme 3A4 (CYP3A4) inhibitors or moderate CYP3A4 inducers, or potent CYP3A4 inducers
* Known hypersensitivity to the IP (active substance or excipients)
* Any other condition or therapy which would make the patient unsuitable for this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 2024-07-09 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Clinical benefit | 6 months
  Hierarchical composite of the following:
  * Time to all-cause mortality
  * Number of total HF events
  * Time to first HF event
  * Difference of 5 points or greater on the Kansas City Cardiomyopathy Questionnaire - Total Symptom Score (KCCQ-TSS) assessed by the win-ratio method
Number of serious adverse events (AEs). | 6 months
  - Serious AEs (excluding efficacy endpoints).
Number of adverse events leading to discontinuation of study drug. | 6 months
  - AEs leading to discontinuation of finerenone or empagliflozin.

SECONDARY OUTCOMES:
Time to first death from any cause or HF event. | 6 months
  Time to first occurrence of all-cause mortality or HF event (hospitalization for HF or urgent visit due to HF)
Mean change from baseline to 6 months in the Total Symptom Score of the Kansas City Cardiomyopathy Questionnaire (KCCQ-TSS). | 6 months
Number of HF events from baseline to Day 90. | 90 days
  - Total (first and recurrent) HF events.

CONTACTS AND LOCATIONS:
Locations (15):
- United States (8):
  - CON-10004 Fairhope, AL Investigational Site, Fairhope, Alabama
  - CON-10075 El Centro, CA Investigational Site, El Centro, California
  - CON-10024 Sacramento, CA Investigational Site, Sacramento, California
  - CON-10022 Atlanta, GA Investigational Site, Atlanta, Georgia
  - CON-10030 Baton Rouge, LA Investigational Site, Baton Rouge, Louisiana
  - CON-10002 Kansas City, MO Investigative Site, Kansas City, Missouri
  - CON-10045 Amarillo, TX Investigational Site, Amarillo, Texas
  - CON-10015 Austin, TX Investigational Site, Austin, Texas
- Brazil (4):
  - CON-21003 Goiania, Goias Investigational Site, Goiânia, Goiás
  - CON-21007 Joinville, Santa Catarina Investigational Site, Joinville, Santa Catarina
  - CON-21004 Braganca Paulista, Sao Paulo Investigational Site, Bragança Paulista, São Paulo
  - CON-21049 Sao Paulo, Sao Paulo Investigational Site, São Paulo, São Paulo
- Canada (3):
  - CON-11012 Surry, BC Investigational Site, Surrey, British Columbia
  - CON-11007 North York, ON Investigational Site, North York, Ontario
  - CON-11005 Sherbrooke, QC Investigational Site, Sherbrooke, Quebec

IPD SHARING:
Plan to Share IPD: No
No current plan to share individual patient data with other researchers.